CLINICAL TRIAL: NCT02466035
Title: Epigenetic Effects Involved in Children With Cow's Milk Allergy: A Possible Effect of Atopic March of Lactobacillus GG (EPICMA)
Brief Title: Epigenetic Effects Involved in Children With Cow's Milk Allergy (EPICMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2815
Record Dates: First submitted 2015-05-27; First posted 2015-06-09 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

ARMS (2):
- Lactobacillus GG (Experimental): Treatment with Lactobacillus rhamnosus GG
  Interventions: Dietary Supplement: Extensively hydrolyzed casein formula plus Lactobacillus rhamnosus GG
- Other formula (No Intervention): Children assuming other hypoallergenic formulas

INTERVENTIONS:
Dietary Supplement: Extensively hydrolyzed casein formula plus Lactobacillus rhamnosus GG — Extensively hydrolyzed casein formula containing the probiotic Lactobacillus rhamnosus GG
  Arms: Lactobacillus GG

SUMMARY:
Lactobacillus GG (LGG) is able to exert long lasting effects in children with atopic disorders. Nutramigen LGG accelerates tolerance acquisition in infants with cow's milk allergy. The mechanisms of these effects are still largely undefined. The effect of LGG could be related at least in part by the immunoregulatory role played by LGG. This probiotic can balance the generation of cytokines possibly involved in IgE- or non-IgE-mediated cow's milk allergy Interleulkin (IL)-4, IL-5, IL-10, IFN-γ , TGF-β, and TNF-Υ), which can contribute to modulation of inﬂammatory processes. The investigators have demonstrated that children with IgE-mediated CMA produce significantly higher level of IL-4 and IL-13 in response to cow's milk protein, and that tolerance is associated with a marked reduction of IL-13 production and a concomitant increased frequency of IFN-γ releasing cells.

Epigenetics studies the heritable (and potentially reversible) changes of the genome inherited from one cell generation to the next which alter gene expression but do not involve changes in primary DNA sequences, highlighting the complexity of the inter-relationship between genetics and nutrition. There are three distinct, but closely interacting, epigenetic mechanisms (histone acetylation, DNA methylation, and non-coding microRNAs) that are responsible for modifying the expression of critical genes associated with physiologic and pathologic processes. The profile of epigenetic modifications associated with Th lineage commitment, coupled with the sensitivity of the early developmental period, has led to speculation that factors that disrupt these pathways may increase the risk of allergic diseases. Specifically, effects on DNA methylation and endogenous histone deacetylase inhibitors acting on specific pathways (Th1 and T regulatory cell differentiation) may favour Th2-associated allergic differentiation. MicroRNAs are another structural components of an epigenetic mechanism of post-transcriptional regulation of messenger RNA translation. It has been recently identified a specific Th2-associated microRNA (miR-21) that is critical for the regulation of Th cell polarization. It has been previously demonstrated an inverse DNA methylation pattern of cytokines involved in Th2 response (IL-4, IL-5) compared with cytokines involved in Th1 response (IL-10, INF- y) in children with CMA acquiring oral tolerance, with the most pronounced effects in those treated with Nutramigen LGG. The current study will prospectively evaluate the effect of Nutramigen LGG and other commercially available hypoallergenic formulas on epigenetic mechanisms that may be related to tolerance acquisition.

ELIGIBILITY:
Inclusion Criteria:

children with cow's milk allergy

Exclusion Criteria:

* Concomitant chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal tract,
* suspected eosinophilic esophagitis or eosinophilic enterocolitis,
* suspected food-protein-induced enterocolitis syndrome,
* suspected cow's milk protein-induced anaphylaxis,
* still on exclusion diet with one of the study formulas or with another dietary regimen because of cow's milk allergy,
* other food allergies.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Epigenetic modifications in cytokines genes | 12 months
  Serum levels (pg/ml) of interleukin 4, interleukin 5, interleukin 10, interferon gamma, FOXP3 in children with cow's milk allergy
Epigenetic modifications in cytokines genes | 12 months
  Methylation rate (%) of interleukin 4, interleukin 5, interleukin 10, interferon gamma, FOXP3 in children with cow's milk allergy

SECONDARY OUTCOMES:
microRNAs modifications | 12 months
  Expression of miR106a, miR126, miR21, miR145, miR27a, miR29a/b, miR155, miR146a, miR128

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy